CLINICAL TRIAL: NCT04990947
Title: Direct Measurement of Food Intake Behaviour in Obese Women Before and After Bariatric Surgery or Lifestyle Intervention
Acronym: CIBuS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1594
Record Dates: First submitted 2021-07-23; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-02

CONDITIONS: Bariatric Surgery Candidate; Lifestyle; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bariatric surgery (Roux-en-Y Gastric Bypass): Patients who are eligible for RYGB
  Interventions: Other: lifestyle / RYGB
- Lifestyle group: Patients with a BMI > 30 who will start a lifestyle program
  Interventions: Other: lifestyle / RYGB

INTERVENTIONS:
Other: lifestyle / RYGB — No intervention, just 2 different groups will be included

SUMMARY:
To assess changes in food intake and food preference (e.g., fat and sugar) after bariatric surgery and lifestyle intervention alone with a direct measurement.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Age between 18 and 67 years of age (standard for eligibility for bariatric surgery)
* Patients must be able to adhere to the study visit schedule
* Independently mobile
* Patients must be able to give informed consent (IC) prior to any study procedures
* Surgical (1) and non-surgical (2) groups:

  1. Eligible for bariatric surgery (BMI > 35 kg/m2 and clinically indicated bariatric surgery operation in agreement with the IFSO criteria)
  2. Patients with a BMI of 30-40 kg/m2, who are planning to join the COOL-lifestyle program

Exclusion Criteria:

* Pre-operatively/lifestyle group: Factors impairing ability to consume meal such as: Significant dysphagia; Gastric outlet obstruction; Anything factor that prevents subjects from drinking or eating a meal
* Post-operatively: Factors impairing ability to consume meal such as: Significant and persistent surgical complications or anything that prevents subjects from drinking or eating a meal.
* Systemic or gastrointestinal condition which may affect food intake or preference (including diabetes mellitus)
* Pregnancy or lactation, or planning to get pregnant during the study period
* Patients who have an intolerance or allergy for one of the components of the test product (e.g. lactose)
* Active and significant psychiatric illness including substance misuse
* Significant cognitive or communication issues
* Medications with documented effect on food intake or food preference
* Participating in another scientific study at the same time, if

Ages: 18 Years to 67 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: RYGB or obesity with lifestyle intervention
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in caloric intake | Before RYGB / lifestyle compared to 4 weeks, 3 months, 6 months and 12 months after RYGB / lifestyle
  kcal consumed

SECONDARY OUTCOMES:
Weight / BMI | baseline, 4weeks, 3 months, 6 months, 12 months
  weight and height measurements
Drinking microstructure over time | baseline, 4weeks, 3 months, 6 months, 12 months
  Measured with the drinkometer
Change in self-reported hunger, thirst, fullness, preference | baseline, 4weeks, 3 months, 6 months, 12 months
  VAS scale 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Yonta van der Burgh, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided